CLINICAL TRIAL: NCT04693637
Title: Phase 2/3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety and Efficacy of ALVR105 (Viralym-M) Compared to Placebo for the Prevention of AdV, BKV, CMV, EBV, HHV-6, and JCV Infection and/or Disease, in High-Risk Patients After Allogeneic Hematopoietic Cell Transplant
Brief Title: Posoleucel (ALVR105, Formerly Viralym-M) for Multi-Virus Prevention in Patients Post-Allogeneic Hematopoietic Cell Transplant
Acronym: Prevent
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AlloVir (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P-105-202 Phase 2
Record Dates: First submitted 2020-12-09; First posted 2021-01-05 (Actual); Results first posted 2024-05-07 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Adenovirus Infection; BK Virus Infection; Cytomegalovirus Infections; Epstein-Barr Virus Infections; Human Herpes Virus-6 Infection; JC Virus Infection
Keywords: Allogeneic Hematopoietic Cell Transplant; Posoleucel; ALVR105; Viralym-M
MeSH Terms: conditions — Adenoviridae Infections; Cytomegalovirus Infections; Epstein-Barr Virus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Posoleucel (ALVR105) (Experimental): Administered as 2-4 milliliter infusion
  Interventions: Biological: Posoleucel (ALVR105)

INTERVENTIONS:
Biological: Posoleucel (ALVR105) — Administered as 2-4 milliliter infusion

SUMMARY:
This is a Phase 2 study to evaluate posoleucel (ALVR105, formerly Viralym-M); an allogeneic, off-the-shelf multi-virus specific T cell therapy that targets six viral pathogens: BK virus, cytomegalovirus, adenovirus, Epstein-Barr virus, human herpesvirus 6 and JC virus.

DETAILED DESCRIPTION:
This is a Phase 2/3, multicenter, randomized, double-blind, placebo controlled trial comparing posoleucel to placebo for the prevention of infection or disease due to AdV, BKV, CMV, EBV, HHV-6, or JCV in high-risk adult and pediatric patients after allogeneic HCT.

There are 2 parts to the study, an open label Phase 2 cohort described in this posting, and a randomized, placebo controlled Phase 3 cohort described in NCT05305040. In the Phase 2 part, 25 to 35 eligible allogeneic HCT recipients will be enrolled and will receive 7 doses of posoleucel over 12 weeks, followed by a 14 week follow-up period.

ELIGIBILITY:
Key Inclusion Criteria

* ≥1 year of age at the day of screening visit.
* Either no evidence of viral infection or viremia, or asymptomatic, viral infection with 3 or fewer viruses of interest at time of screening
* Within 15 and 42 days of receiving a first allogeneic HCT and have demonstrated clinical engraftment
* Meet one or more of the following criteria at the time of randomization:

  * Related (sibling) donor with at least one mismatch at one of these HLA-gene loci: HLA-A, -B or -DR
  * Haploidentical donor
  * Unrelated donor with at least one mismatch at one of these HLA-gene loci: HLA-A, -B, -C, or -DR
  * Use of umbilical cord blood as stem cell source
  * Ex vivo graft manipulation resulting in T cell depletion
  * Lymphocyte Count <180/mm3 and/or cluster of differentiation 4 (CD4) Count <50/mm3

Key Exclusion Criteria:

* History of AdV, BKV, CMV, EBV, HHV-6, and/or JCV end-organ disease within 6 months prior to randomization
* Evidence of active Grade >2 acute GVHD
* Presence of non-minor uncontrolled or progressive bacterial, viral or fungal infections
* Known history or current (suspected) diagnosis of CRS requiring treatment associated with the administration of peptides, proteins, and/or antibodies
* Ongoing therapy with high-dose systemic corticosteroids (ie, prednisone equivalent dose >0.5 mg/kg/day) within 24 hours prior to dosing
* Relapse of primary malignancy other than minimal residual disease

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-01-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope National Medical Center, Duarte, California
  - University of California, San Francisco Medical Center, San Francisco, California
  - Childrens National Medical Center, Northwest Rectangle, District of Columbia
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Kansas Hospital, Westwood, Kansas
  - University of Maryland Medical Center, Baltimore, Maryland
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - Children's Mercy Kansas City, Kansas City, Missouri
  - Weill Cornell Medical College, New York, New York
  - Stony Brook University Hospital Cancer Center, Stony Brook, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Medical Center Dallas, Dallas, Texas
  - University of Virginia, Charlottesville, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Posoleucel (ALVR105), an Off-the-Shelf, Multivirus-Specific T-Cell Therapy, for the Prevention of Viral Infections Post-HCT: Results from an Open-Label Cohort of a Phase 2 Trial Sanjeet S Dadwal, Michael Shuster, Gary Douglas Myers, Keith Boundy, Marshelle Warren, Elizabeth Stoner, Thuy Truong, Joshua A. Hill Blood (2021) 138 (Supplement 1): 1760.
- [Background] Tzannou I, Papadopoulou A, Naik S, Leung K, Martinez CA, Ramos CA, Carrum G, Sasa G, Lulla P, Watanabe A, Kuvalekar M, Gee AP, Wu MF, Liu H, Grilley BJ, Krance RA, Gottschalk S, Brenner MK, Rooney CM, Heslop HE, Leen AM, Omer B. Off-the-Shelf Virus-Specific T Cells to Treat BK Virus, Human Herpesvirus 6, Cytomegalovirus, Epstein-Barr Virus, and Adenovirus Infections After Allogeneic Hematopoietic Stem-Cell Transplantation. J Clin Oncol. 2017 Nov 1;35(31):3547-3557. doi: 10.1200/JCO.2017.73.0655. Epub 2017 Aug 7. PMID 28783452
- [Background] Chandraker A, Regmi A, Gohh R, Sharma A, Woodle ES, Ansari MJ, Nair V, Chen LX, Alhamad T, Norman S, Cibrik D, Singh M, Alper A, Jain D, Zaky Z, Knechtle S, Sharfuddin A, Gupta G, Lonze BE, Young JH, Adey D, Faravardeh A, Dadhania DM, Rossi AP, Florescu D, Cardarelli F, Ma J, Gilmore S, Vasileiou S, Jindra PT, Wojciechowski D. Posoleucel in Kidney Transplant Recipients with BK Viremia: Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase 2 Trial. J Am Soc Nephrol. 2024 May 1;35(5):618-629. doi: 10.1681/ASN.0000000000000329. Epub 2024 Mar 12. PMID 38470444
- [Derived] Dadwal SS, Bansal R, Schuster MW, Yared JA, Myers GD, Matzko M, Adnan S, McNeel D, Ma J, Gilmore SA, Vasileiou S, Leen AM, Hill JA, Young JH. Final outcomes from a phase 2 trial of posoleucel in allogeneic hematopoietic cell transplant recipients. Blood Adv. 2024 Sep 10;8(17):4740-4750. doi: 10.1182/bloodadvances.2023011562. PMID 38593233

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Posoleucel (ALVR105)
Started | 26
Completed | 16
Not Completed | 10
Not completed — Death | 4
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Analysis Population will include all patients who received posoleucel.
Arm/Group | Posoleucel (ALVR105)
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 17
  >=65 years | 8
Age, Continuous [Median (Full Range); unit: years] | 59.5 [14 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 18
  More than one race | 3
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26
Underlying Disease [Count of Participants; unit: Participants]
  Leukemia | 17
  Myelodysplasia/Myeloproliferative | 3
  Lymphoma | 2
  Sickle Cell Anemia | 2
  Other | 2
Type of Transplant [Count of Participants; unit: Participants]
  Haploidentical | 12
  Mismatched Unrelated | 9
  Matched Unrelated | 4
  Umbilical Cord Blood | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Clinically Significant Infections or Episodes of End-organ Disease
Description: The number of participants experiencing clinically significant infections or episodes of end-organ disease due to AdV, BKV, CMV, EBV, HHV-6, or JCV through Week 14
Time Frame: Through Week 14
Measure: Count of Participants; unit: Participants
Arm/Group | Posoleucel (ALVR105)
Number analyzed (Participants) | 26
Participants | 3

2. Secondary Outcome: Number of Participants Experiencing Clinically Significant Infections or Episodes of End-organ Disease
Description: The number of participants experiencing clinically significant infections or episodes of end-organ disease due to AdV, BKV, CMV, EBV, HHV-6, or JCV through Week 26.
Time Frame: Through Week 26
Measure: Count of Participants; unit: Participants
Arm/Group | Posoleucel (ALVR105)
Number analyzed (Participants) | 26
Participants | 7

3. Secondary Outcome: Number of Participants Experiencing Clinically Significant Infections or Episodes of End-organ Disease Due to Adenovirus (AdV)
Description: The number of participants experiencing clinically significant infections or episodes of end-organ disease due to AdV, BKV, CMV, EBV, HHV-6, or JCV from each individual virus through Week 26 (6 endpoints each at Week 26).
Time Frame: Through Week 26
Measure: Count of Participants; unit: Participants
Arm/Group | Posoleucel (ALVR105)
Number analyzed (Participants) | 26
Participants | 1

4. Secondary Outcome: Number of Participants Experiencing Clinically Significant Infections or Episodes of End-organ Disease Due to BKV
Description: The number of participants experiencing clinically significant infections or episodes of end-organ disease due to AdV, BKV, CMV, EBV, HHV-6, or JCV from each individual virus through Week 14 and Week 26 (6 endpoints each at Week 14 and Week 26).
Time Frame: Through Week 26
Measure: Count of Participants; unit: Participants
Arm/Group | Posoleucel (ALVR105)
Number analyzed (Participants) | 26
Participants | 0

5. Secondary Outcome: Number of Participants Experiencing Clinically Significant Infections or Episodes of End-organ Disease Due to Cytomegalovirus (CMV)
Description: as for outcome 3
Time Frame: Through Week 26
Measure: Count of Participants; unit: Participants
Arm/Group | Posoleucel (ALVR105)
Number analyzed (Participants) | 26
Participants | 5

6. Secondary Outcome: Number of Participants Experiencing Clinically Significant Infections or Episodes of End-organ Disease Due to Epstein-Barr Virus (EBV)
Description: as for outcome 3
Time Frame: through Week 26
Measure: Count of Participants; unit: Participants
Arm/Group | Posoleucel (ALVR105)
Number analyzed (Participants) | 26
Participants | 1

7. Secondary Outcome: Number of Participants Experiencing Clinically Significant Infections or Episodes of End-organ Disease Due to Human Herpes Virus 6 (HHV-6)
Description: as for outcome 3
Time Frame: Through Week 26
Measure: Count of Participants; unit: Participants
Arm/Group | Posoleucel (ALVR105)
Number analyzed (Participants) | 26
Participants | 0

8. Secondary Outcome: Number of Participants Experiencing Clinically Significant Infections or Episodes of End-organ Disease Due to John Cunningham Virus (JCV)
Description: as for outcome 3
Time Frame: Through Week 26
Measure: Count of Participants; unit: Participants
Arm/Group | Posoleucel (ALVR105)
Number analyzed (Participants) | 26
Participants | 0

9. Secondary Outcome: Rates of Overall and Non-Relapse Mortality
Description: The number of mortality events due to non-relapse causes through Week 52.
Time Frame: Through Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | Posoleucel (ALVR105)
Number analyzed (Participants) | 26
Participants
  Overall Mortality | 4
  Non-Relapse Mortality | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed up to week 52; serious and other (not including serious) adverse events were assessed for up to week 26
Arm/Group | Posoleucel (ALVR105)
All-Cause Mortality (participants affected / at risk) | 4/26
Serious Adverse Events (participants affected / at risk) | 19/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Posoleucel (ALVR105) (N=26)
Adrenoleukodystrophy (Congenital, familial and genetic disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Pancreatitis Acute (Gastrointestinal disorders) | 1
Pancreatitis Necrotising (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 2
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 2
Acute graft versus host disease in skin (Immune system disorders) | 1
Chronic graft versus host disease in lung (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Sepsis (Infections and infestations) | 3
Cytomegalovirus infection reactivation (Infections and infestations) | 2
Adenovirus infection (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
COVID 19 (Infections and infestations) | 1
Enterocolitis bacterial (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Genital herpes simplex (Infections and infestations) | 1
Klebsiella bacteraemia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Transplant Failure (Injury, poisoning and procedural complications) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute Myeloid Leukemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Post Transplant Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Seizure (Nervous system disorders) | 1
Mental Disorder (Psychiatric disorders) | 1
Suicidal Ideation (Psychiatric disorders) | 1
Acute Kidney injury (Renal and urinary disorders) | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 1
Nephrotic syndrome (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Posoleucel (ALVR105) (N=26)
Anaemia (Blood and lymphatic system disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 16
Abdominal Pain (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 4
Abdominal Pain Lower (Gastrointestinal disorders) | 2
Abdominal tenderness (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 2
Chills (General disorders) | 5
Fatigue (General disorders) | 5
Oedema peripheral (General disorders) | 4
Pain (General disorders) | 4
Pyrexia (General disorders) | 4
Catheter site pain (General disorders) | 2
Acute graft versus host disease in skin (Immune system disorders) | 10
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 3
Chronic graft versus host disease in skin (Immune system disorders) | 2
Chronic graft versus host disease oral (Immune system disorders) | 2
Cytomegalovirus infection reactivation (Infections and infestations) | 3
Cytomegalovirus viraemia (Infections and infestations) | 3
Sepsis (Infections and infestations) | 3
Urinary Tract infection (Infections and infestations) | 3
COVID-19 (Infections and infestations) | 2
Polyomavirus viraemia (Infections and infestations) | 2
Upper Respiratory tract infection (Infections and infestations) | 2
Procedural Pain (Injury, poisoning and procedural complications) | 2
Transplant Failure (Injury, poisoning and procedural complications) | 2
Weight decreased (Investigations) | 6
Platelet count decreased (Investigations) | 5
Blood creatinine increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 3
White blood cell count decreased (Investigations) | 3
Alanine aminotransferase increased (Investigations) | 2
Decreased Appetite (Metabolism and nutrition disorders) | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2
Tremor (Nervous system disorders) | 6
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 4
Presyncope (Nervous system disorders) | 2
Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 2
Acute Kidney injury (Renal and urinary disorders) | 2
Pollakiuria (Renal and urinary disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 3
Erythema (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Skin Lesion (Skin and subcutaneous tissue disorders) | 2
Hypotension (Vascular disorders) | 3
Hypertension (Vascular disorders) | 2
Dry eye (Eye disorders) | 2
Photophobia (Eye disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-04-07): https://cdn.clinicaltrials.gov/large-docs/37/NCT04693637/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-30): https://cdn.clinicaltrials.gov/large-docs/37/NCT04693637/SAP_001.pdf